CLINICAL TRIAL: NCT05000398
Title: Comparison of the Effects of Advanced Exercise Treatment Performed Under the Supervision of a Physiotherapist and Provided as a Home Program on Adduction Angle, Pain, Functional Status, Quality of Life and Kinesophobia in Individuals With Hallux Valgus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Merve Betül Öztarsu, physiotherapist, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMerve
Record Dates: First submitted 2021-08-08; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Exercise; Hallux Valgus
Keywords: hallux valgus; exercise; home program
MeSH Terms: conditions — Motor Activity; Hallux Valgus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise with a physiotherapist (Active Comparator): Participants will exercise with a physiotherapist. 4 times a week for 8 weeks
  Interventions: Other: Stretching the intrinsic muscles; Other: Thumb Abduction with MTF Joint Traction; Other: Thumb active extension exercise; Other: Toe spread out; Other: Short foot; Other: Heel rise; Other: Towel toe curl; Other: Gastrocnemius active static stretching exercise; Other: Plantar fascia and gastrocnemius stretching exercise on step
- home program (Experimental): The same exercises will be given to the participants as brochures. 4 times a week for 8 weeks
  Interventions: Other: Stretching the intrinsic muscles; Other: Thumb Abduction with MTF Joint Traction; Other: Thumb active extension exercise; Other: Toe spread out; Other: Short foot; Other: Heel rise; Other: Towel toe curl; Other: Gastrocnemius active static stretching exercise; Other: Plantar fascia and gastrocnemius stretching exercise on step

INTERVENTIONS:
Other: Stretching the intrinsic muscles — Participants will be asked to dorsiflex the foot and stretch for 30 seconds. It will be done with 5 repetitions.
Other: Thumb Abduction with MTF Joint Traction — participants will be held for 30 seconds by passively abducting the thumb within the limits of pain, and will be applied with 5 repetitions.
Other: Thumb active extension exercise — An elastic band will be placed around the thumb, stretching enough to ensure proper alignment of the thumb and passively correct the position. It will be desired to move the feet away from each other without moving the heels from the ground and the extension movement of the thumbs.2 sets will be performed as 10 repetitions. 30 seconds of rest will be given to prevent fatigue between sets.
Other: Toe spread out — In the first stage, active finger extension and abduction will be requested while the heel and metatarsal heads are in contact with the ground. In the second stage, while the other fingers are in extension, the smallest finger will be brought laterally and flexed to contact the ground. In the third stage, while in the second stage position, the thumb will be brought into abduction and flexion slowly and contact with the ground will be requested. These 3 phases will be repeated sequentially.2 sets will be performed as 10 repetitions. 30 seconds of rest will be given to prevent fatigue between sets.
Other: Short foot — While standing , the medial arch will be raised by trying to bring the metatarsal heads closer to the heel . The patient will be asked to move the big toe closer to the heel without bending the toes and without lifting the heel off the ground.2 sets will be performed as 10 repetitions. 30 seconds of rest will be given to prevent fatigue between sets.
Other: Heel rise — After taking a 5 cm high tape measure against the wall, the person will be asked to stand up on her heel by at least 5 cm.2 sets will be performed as 10 repetitions. 30 seconds of rest will be given to prevent fatigue between sets.
Other: Towel toe curl — Patients will be asked to place their feet on the edge of the towel on the floor. An elastic band will be placed around the thumb, stretching enough to ensure proper alignment of the thumb and passively correct the position. Next, they will be asked to grasp the towel with their fingers, flexing their toes, and forcefully dragging them under their feet.2 sets will be performed as 10 repetitions. 30 seconds of rest will be given to prevent fatigue between sets.
Other: Gastrocnemius active static stretching exercise — The patient will be placed on the wall at eye level, 50 centimeters away from the wall. The leg that is desired to be stretched will be brought back, while the knee is straight, it will be requested to flex the front leg. During the test, it will be requested that the back heel does not rise from the ground and wait 30 seconds. 5 repetitions to be done
Other: Plantar fascia and gastrocnemius stretching exercise on step — The patient will be asked to place both feet on the step and slowly stretch the heel downwards until a stretch is felt in the arch of the foot and wait 30 seconds. 5 repetitions will be done

SUMMARY:
The aim of our study is to compare the effects of progressive exercise therapy, administered as a home program under the supervision of a physiotherapist, on adduction angle, pain, functional status, quality of life, and kinesiophobia in individuals aged 18-64 years with a hallux valgus angle of 15-40 degrees (mild-moderate).

DETAILED DESCRIPTION:
According to the power analysis, 18 people will participate in the study. Individuals with halluk valgus pain, deformity angle, balance, functional capacity, functionality, quality of life and kinesiophobia will be evaluated.After the individuals are evaluated, they will be randomly divided into 2 groups as the exercise group and the home exercise group.

All patients will be instructed on wearing appropriate footwear (made of soft material, with a wide round toe, with a normal heel height between 1 inch and 1.5 inches (2.5-3.8 cm). In addition, in order to increase the awareness of the participants, they will be asked to focus on how muscle activation feels during exercise and they will be asked to perform this activation during daily living activities.

The exercise program to be given to both groups will be the same, and will be applied with bare feet 4 days a week for 8 weeks. The exercise program will be advanced as recommended in the literature and 30 seconds of rest will be given between sets.

After the evaluation, all exercises will be shown to the home exercise group and it will be ensured that they are applied correctly. An illustrated and narrative exercise program brochure containing information about exercise position, number of repetitions, contraction time, rest time between sets, frequency and exercise diary will be given to the patient for exercise follow-up.

At the end of 8 weeks, the evaluations will be repeated by the same physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer individuals between the ages of 18-64
* Mild to moderate (15-40 degrees) hallux valgus
* Bilateral hallux valgus
* Have not received physical therapy for hallux valgus in the last 6 months,
* Individuals who did not use orthotic devices or dynamic splints for the treatment of hallux valgus will be included in the study.

Exclusion Criteria:

* HVA ≥ 45°
* Rjjit hallux valgus deformity (in cases where the hallux cannot be brought to its normal position manually)
* Obesity (BMI>30 kg/m2)
* Systemic disease and inflammatory arthritis (rheumatoid arthritis, systemic lupus, diabetes mellitus)
* Neurological disease (eg: neuropathy)
* Vestibular disorder that may affect balance
* History of standing trauma, fracture of the metatarophalangeal joint,
* He has undergone foot-ankle surgery,
* Using NSAIDs or analgesics

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-08-16 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
hallux valgus angle | Change from Baseline and at the end of 8 weeks
  The hallux valgus angle will be measured with a goniometer at the beginning and end of the treatment.

SECONDARY OUTCOMES:
hallux valgus pain | Change from Baseline and at the end of 8 weeks
  Hallux valgus pain will be measured with the VAS scale at the beginning and end of treatment.
Functional Status | Change from Baseline and at the end of 8 weeks
  Static Balance Evaluation: It will be evaluated with the one-leg standing test.Dynamic Balance Evaluation: It will be evaluated by Y balance test.Functional capacity: To be evaluated with a 6-minute walk test.Foot Function Index (FFI): This index measures pain, function and activity limitation
life quality | Change from Baseline and at the end of 8 weeks
  The SF-36 quality of life questionnaire will be used to assess general health-related quality of life.
kinesiophobia | Change from Baseline and at the end of 8 weeks
  The Tampa Kinesiophobia Scale will be used to measure the fear of movement or re-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Öksüz, assist.prof., Study Director — Eastern Mediterranean University
Locations (1):
- Merve Betül Öztarsu, Famagusta, Cyprus